CLINICAL TRIAL: NCT04815733
Title: Pressure Support Ventilation During Laparoscopic and Abdominal Robotic Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Principal Investigator, Valerii Subbotin, PhD, Moscow Clinical Scientific Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MoscowCSC
Record Dates: First submitted 2020-10-28; First posted 2021-03-25 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Ventilator-Induced Lung Injury
Keywords: pressure support ventilation; anaesthesia; lung injury; laparoscopic surgery
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Lung Injury

STUDY DESIGN:
Intervention Model Description: t is planned to recruit patients in two groups: group 1-patients who will undergo General anesthesia with deep neuromuscular block and PCV-VG; group 2-patients with partial neuromuscular block and PSVpro.
  Randomization of patients into two 1:1 groups will be performed by random number generation.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandatory ventilation (Active Comparator): deep neuromuscular block and mandatory ventilation (PCV-VG);
  Interventions: Procedure: Mandatory ventilation
- Pressure support ventilation (Experimental): partial neuromuscular block and pressure support ventilation (PSVpro).
  Interventions: Procedure: pressure support ventilation

INTERVENTIONS:
Procedure: Mandatory ventilation — Use PCV-VG
  Arms: Mandatory ventilation
Procedure: pressure support ventilation — Use PSVpro
  Arms: Pressure support ventilation

SUMMARY:
This study is a single-center, blind, prospective, randomized, controlled trial of pressure support ventilation (PSVpro) versus pressure control ventilation - volume guaranteed (PCV - VG) during laparoscopic and robotic abdominal surgery.

DETAILED DESCRIPTION:
The objective of the study to evaluate the possibility and feasibility of using PSVpro during anesthesia during long-term laparoscopic and robot-assisted abdominal operations at different levels of neuromuscular block.

Intervention: We plan to include 100 patients who will undergo elective long (more 2 hours) laparoscopic or abdominal robotic surgery. All patients will be randomly assigned in two groups in ratio 1:1. 1 group- deep neuromuscular block and mandatory ventilation; 2 group- partial neuromuscular block and pressure support ventilation.

Expected Results. PSV may reduce the systemic inflammatory response compared to the mandatory ventilation during laparoscopic and abdominal robotic surgery.

ELIGIBILITY:
Inclusion criteria:

* Written consent.
* Men and women aged 18 years or more.
* The physical status from ASA classification I, II or III.
* BMI <= 34.9 kg / m2.
* Low risk of respiratory complications.
* Laparoscopic surgery in the pelvis.

Exclusion criteria:

* The physical status from ASA IV or V.
* BMI> = 35 kg / m2.
* Neuromuscular disease.
* Allergy to Anesthetic Agents.
* Operations on two cavities.
* Operations on the chest cavity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Concentrations of biomarkers of lung injury | 1-3 hours after surgery
  Measure concentration of Interleukin-6 (IL-6), Interleukin-8 (IL-8), tumor necrosis factor receptor I / II (sTNF rI / II)) in blood serum

SECONDARY OUTCOMES:
Maximum intraoperative lactate level in the early postoperative period | 1 hour after surgery
  Maximum intraoperative lactate level
The maximum level of vasopressor support during surgery | From time of skin incision to time of skin closure assessed up to 24 hours
  Norepinephrine consumption (mcg/kg/h)

OTHER OUTCOMES:
Duration of anaesthesia. | Period of time from induction to volatile anesthetic supply stop assessed up to 24 hours
  Duration of anaesthesia.
Procedure time | Period of time from intubation to extubation assessed up to 24 hours
  Length of ventilation
Length of stay (LOS) in the intensive care unit (ICU). | Period of time from ICU arrival to discharge from ICU assessed up to 1 year
  Length of stay (LOS) in the intensive care unit (ICU).
Time to reach an Aldrete score > 9 points after anaesthesia | Period of time from volatile anesthetic suplly stop to time when patient has more than 9 points according Aldrete score assessed up to 24 hours
  Time to reach an Aldrete score > 9 points after anaesthesia
Intraoperative consumption of muscle relaxant | Since skin incision to skin closure assessed up to 24 hours
  mg/kg of muscle relaxant
Intraoperative consumption of reversal agents. | Since skin incision to skin closure assessed up to 24 hours
  mg/kg of reversal agents.
Supplemental oxygen in the early postoperative period | Since extubation up to 24 hours after extubation
  Duration of oxygen supply
Quality of recovery score-40 | 24 hours after surgery
  The QoR-40 incorporates five dimensions of health: patient support, comfort, emotions, physical independence, and pain; each item is graded on a five-point Likert scale.
  QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Changes of spirometry parameter FVC after surgery | 1 hour and 24 hours after surgery
  FVC before surgery (L) - FVC after surgery (L)
Changes of spirometry parameter FEV1 after surgery | 1 hour and 24 hours after surgery
  FEV1 before surgery (L)- FEV1 after surgery (L)
Changes of spirometry parameter FEV1/FVC after surgery | 1 hour and 24 hours after surgery
  FEV1/FVC before surgery (percentage %) - FEV1/FVC after surgery (percentage %)
Changes of spirometry parameter PEF after surgery | 1 hour and 24 hours after surgery
  PEF before surgery (L/s) - PEF after surgery (L/s)
Changes of spirometry parameter VC after surgery | 1 hour and 24 hours after surgery
  VC before surgery (L) - VC after surgery (L)
Changes of spirometry parameter FEV1/VC after surgery | 1 hour and 24 hours after surgery
  FEV1/VC before surgery (percentage %) - FEV1/VC after surgery (percentage %)
Volume of atelectasis of lungs after surgery | 24 hours after surgery
  Volume of the lungs measure according to CT lung The volume of atelectasis is the difference in volumes of lungs before and after surgery
The level of pain assess after surgery by Numeric Rating Scale (NRS) | 1 hour after surgery
  No pain - 0, worst pain - 10
The level of pain assess after surgery by Numeric Rating Scale (NRS) | 3 hours after surgery
  No pain - 0, worst pain - 10
The level of pain assess after surgery by Numeric Rating Scale (NRS) | 24 hours after surgery
  No pain - 0, worst pain - 10
Length of stay (LOS) in hospital | 28 days
  Length of stay (LOS) in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow Clinical Scientific Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No